CLINICAL TRIAL: NCT06169072
Title: Sentinel Lymph Node Localisation With an Ultra-low Dose of Superparamagnetic Iron Oxide Nanoparticles in Patients With Breast Cancer
Brief Title: Sentinel Lymph Node Localisation With an Ultra-low Dose of Magtrace in Breast Cancer Patients
Acronym: MagSnow2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Professor, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SUGBG-2022002
Record Dates: First submitted 2023-11-18; First posted 2023-12-13 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: Breast cancer; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — ferumoxides

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sentinel node detection with 0.1mL SPIO and Technetium99 (Other): An intradermal injection of SPIO (MagTrace®), according to the pre-specified dose of 0.1mL, will be performed 7 days, up to the day of surgery. The injection should be in the skin over the tumour, or at the border of the areola. All patients will also receive technetium per routine.
  Interventions: Drug: Superparamagnetic Iron Oxide; Device: Technetium99

INTERVENTIONS:
Drug: Superparamagnetic Iron Oxide — Superparamagnetic iron oxide (SPIO) consists of an iron oxide nanoparticle core and a hydrophilic coating to make it biocompatible and colloidal stable in a suspension. In this study injected intradermally in an ultra-low dose
  Other Names: Magtrace
Device: Technetium99 — Technetium99 +/- blue dye is injected per routine as a comparator and as back up.

SUMMARY:
The overall aim is to demonstrate that the use of superparamagnetic iron oxide nanoparticles (SPIO) as a tracer in an ultra-low dose (0.1 ml) is non-inferior for sentinel lymph node (SLN) detection in patients with breast cancer compared to the dual technique using Tc99m +/- blue dye, and to evaluate MRI breast artefacts and skin staining over time.

DETAILED DESCRIPTION:
The overall aim is to demonstrate that the use of superparamagnetic iron oxide nanoparticles (SPIO) as a tracer in an ultra-low dose (0.1 ml) is non-inferior for sentinel lymph node (SLN) detection in patients with breast cancer compared to the dual technique using Tc99m +/- blue dye, and to evaluate MRI breast artefacts and skin staining over time.

This is a prospective cohort study where all research persons have SLN biopsy using both SPIO and the dual technique. Then the investigators will compare SLN detection rates between Magtrace 0.1 ml and the dual routine technique with radioactive tracer (Technetium99m, Tc99) +/- blue dye.

ELIGIBILITY:
Inclusion Criteria:

* Planned for sentinel lymph node biopsy at (or after) breast surgery
* Signed and dated written informed consent before the start of specific protocol procedures

Exclusion Criteria:

* Pregnant or breast-feeding
* Iron overload disease
* Known hypersensitivity to iron, dextran compounds or blue dye.
* Inability to understand given information and give informed consent or undergo study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
SLN detection rate for Magtrace 0.1 ml and for dual technique (Tc99 +/- blue dye) measured as per cent of patients where a SLN is identified using either the magnetic or the dual technique. | During the procedure
  percentage

SECONDARY OUTCOMES:
MRI Magtrace artefacts | 3-6, 12 and 24-36 months postoperatively
  Measured as per cent of patients with remaining artefacts evaluated by blinded central review.
Skin staining due to injected Magtrace | 4 weeks, 12, 24 and 36 months postoperatively
  Measured as per cent of patients with remaining brown or blue skin staining and stain size, evaluated by the investigator and the Skin Discoloration Impact Evaluation Questionnaire (SDIEQ)
Rate of device-related AE and SAEs | During the procedure
  Number
Numbers of nodes detected and removed for Magtrace 0.1 ml and for the dual technique (Tc99 +/- blue dye) | During the procedure
  Numbers
Concordance between detected SLN by Magtrace 0.1 ml or by the dual technique (Tc +/- blue dye) | During the procedure
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Wärnberg, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska Iniversity Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balch CM. Detection of melanoma metastases with the sentinel node biopsy: the legacy of Donald L. Morton, MD (1934-2014). Clin Exp Metastasis. 2018 Aug;35(5-6):425-429. doi: 10.1007/s10585-018-9908-8. Epub 2018 May 31. PMID 29855858
- [Background] Waanders S, Visscher M, Wildeboer RR, Oderkerk TO, Krooshoop HJ, Ten Haken B. A handheld SPIO-based sentinel lymph node mapping device using differential magnetometry. Phys Med Biol. 2016 Nov 21;61(22):8120-8134. doi: 10.1088/0031-9155/61/22/8120. Epub 2016 Oct 26. PMID 27782005
- [Background] Karakatsanis A, Daskalakis K, Stalberg P, Olofsson H, Andersson Y, Eriksson S, Bergkvist L, Warnberg F. Superparamagnetic iron oxide nanoparticles as the sole method for sentinel node biopsy detection in patients with breast cancer. Br J Surg. 2017 Nov;104(12):1675-1685. doi: 10.1002/bjs.10606. Epub 2017 Sep 6. PMID 28877348
- [Background] Mirzaei N, Katsarelias D, Zaar P, Jalnefjord O, Johansson I, Leonhardt H, Warnberg F, Olofsson Bagge R. Sentinel lymph node localization and staging with a low-dose of superparamagnetic iron oxide (SPIO) enhanced MRI and magnetometer in patients with cutaneous melanoma of the extremity - The MAGMEN feasibility study. Eur J Surg Oncol. 2022 Feb;48(2):326-332. doi: 10.1016/j.ejso.2021.12.467. Epub 2022 Jan 1. PMID 35000820
- [Background] Karakatsanis A, Christiansen PM, Fischer L, Hedin C, Pistioli L, Sund M, Rasmussen NR, Jornsgard H, Tegnelius D, Eriksson S, Daskalakis K, Warnberg F, Markopoulos CJ, Bergkvist L. The Nordic SentiMag trial: a comparison of super paramagnetic iron oxide (SPIO) nanoparticles versus Tc(99) and patent blue in the detection of sentinel node (SN) in patients with breast cancer and a meta-analysis of earlier studies. Breast Cancer Res Treat. 2016 Jun;157(2):281-294. doi: 10.1007/s10549-016-3809-9. Epub 2016 Apr 27. PMID 27117158
- [Background] Hersi AF, Pistiolis L, Dussan Luberth C, Vikhe-Patil E, Nilsson F, Mohammed I, Olofsson Bagge R, Warnberg F, Eriksson S, Karakatsanis A. Optimizing Dose and Timing in Magnetic Tracer Techniques for Sentinel Lymph Node Detection in Early Breast Cancers: The Prospective Multicenter SentiDose Trial. Cancers (Basel). 2021 Feb 9;13(4):693. doi: 10.3390/cancers13040693. PMID 33572114

DOCUMENTS (1):
  • Study Protocol (2023-02-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT06169072/Prot_000.pdf